CLINICAL TRIAL: NCT02774603
Title: The Efficacy of Aquatic Locomotor Training Compared to Overground Locomotor Training in Improving Ambulatory Function and Health-Related Quality of Life
Brief Title: Aquatic vs. Land Locomotor Training Overground Locomotor Training in Improving Ambulatory Function and Health-Related Quality of Life
Acronym: ALT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to lack of funding the study was terminated early
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Cristina Sadowsky, M.D., Assistant Professor, Director, Physician, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00066544
Record Dates: First submitted 2016-05-12; First posted 2016-05-17 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Aquatic Locomotor Training (Active Comparator): Aquatic Locomotor Training is a Locomotor Training technique utilizing an underwater treadmill to help increase a patient's independence and function. Aquatic Locomotor Training may require up to three people to obtain desirable gait kinematics: one at each of the patient's legs, and one at the patient's pelvis; however, typically with ambulatory patients, only one therapist is utilized. Therapists are highly trained, using their legs and feet to provide properly timed underwater cues throughout the gait cycle.
  Interventions: Other: Aquatic Locomotor Training
- Land Locomotor Training (Active Comparator): Locomotor Training encompasses a variety of interventions ranging from BWSTT to overground gait training to robotic-assisted walk training. Overground Locomotor Training, depending upon the technique used, can require up to four people to complete the intervention (one at each participant's leg, one at the participant's trunk and/or pelvis, and one monitoring the computer and/or treadmill).
  Interventions: Other: Land Locomotor Training

INTERVENTIONS:
Other: Aquatic Locomotor Training
  Arms: Aquatic Locomotor Training
Other: Land Locomotor Training
  Arms: Land Locomotor Training

SUMMARY:
The aim of this study is to define and evaluate the efficacy of Aquatic Locomotor Training (ALT) compared to overground Locomotor Training in improving ambulatory function and health-related quality of life. The investigators hypothesize, that Aquatic Locomotor Training is capable of producing outcomes that are as good as, or better than, overground Locomotor Training.

Aquatic Locomotor Training may be another tool for therapists to utilize for clinical improvements in function and gait for the Spinal Cord Injury (SCI) population.

To determine the efficacy of Aquatic Locomotor Training on improving rehabilitation outcomes among patients with incomplete traumatic cervical Spinal Cord Injury by assessing these parameters:

1. Walking speed and endurance
2. Functional balance and fall risk
3. HRQoL

To describe the feasibility of conducting Aquatic Locomotor Training as an Locomotor Training modality for the rehabilitation of patients with incomplete traumatic cervical Spinal Cord Injury.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-65 years
2. Cervical level (C1-C7) SCI of traumatic origin
3. Motor incomplete SCI (ASIA Impairment Scale C or D)
4. Chronic SCI, >12 months
5. Age between 18 to 65 years
6. Functional Status

i. Overground ambulator (able to walk at least 10 m with or without an assistive device)

ii. Able to demonstrate active movement at/or below L2 myotome

iii. Able to demonstrate adequate head control

1. Voluntarily extend head while positioned in harness

iv. Tolerance to activity

1. Participant able to tolerate up to 1 hour of standing without experiencing symptoms of orthostatic hypotension

g. Range of motion

i. PROM values for ankle dorsiflexion

1. Neutral positioning, 0○

ii. PROM values for knee extension

1. Up to -10○

iii. PROM values for hip extension

1. Neutral positioning, 0○

h. Height

i. Participant with minimum height of 48"

i. Weight

i. Participant with minimum weight of (to be determined based on therapist's clinical judgment)

ii. Participant with maximum weight of 300 lb

j. Participants are able to comply with procedures and follow up

k. Participants are medically stable, with no recent (1 month or less) inpatient admission for acute medical or surgical issues

l. Participants are legally able to make their own health care decisions

Exclusion Criteria:

a. Medical Complications i. Fracture

1. Participant with presence of unhealed fracture ii. Physician hold for medical reasons that the Principle Investigator will judge and decide on a case by case basis as a potential safety threat to the participant

1. Wounds a. Allowed if physician cleared i. Excluded wounds likely to be present in areas enclosed with harness, present in areas that require access for facilitation, present in areas of direct weight bearing during LT session b. Wounds allowed must be fully covered with gauze then opsite (waterproof bandage) before Aquatic Locomotor Training
2. Comorbidities a. E.g. poorly controlled diabetes, uncontrolled seizures, etc.
3. Orthostatic hypotension

   a. Participant demonstrates symptomatic orthostatic hypotension that limits activity
4. Uncontrolled autonomic dysreflexia symptoms a. Episode of uncontrolled autonomic dysreflexia symptoms within the past 1 month iii. Diarrhea iv. Mechanical ventilation v. Pacemakers vi. Central lines vii. Women who are pregnant, confirmed by a urine pregnancy test that will be done on all menstruating, or non-menopausal women viii. History of neurological disease ix. Non English speaking participants will not be targeted b. Currently undergoing, or have received Aquatic Locomotor Training or overground Locomotor Training within four weeks of the study start date (see above in 4d for further details)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Change from Baseline 10 meter Walk Test at 4 months | up to 16 weeks

SECONDARY OUTCOMES:
6 Minute Walk Test | up to 16 weeks
Berg Balance Scale | up to 16 weeks
Health Survey on the Short Form 36 | up to 16 weeks
Quality of Life on the SCI QL-23 scale | up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Sadowsky, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Cristina Sadowsky, M.D., Baltimore, Maryland, United States